CLINICAL TRIAL: NCT06208384
Title: Efficacy and Safety of Topical Statin Eye Drop in the Management of Dry Eye Associated With Meibomian Gland Dysfunction
Brief Title: Topical Statin Eye Drop in the Management of the Dry Eye
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammadali Javadi, MD, Head of Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14023
Record Dates: First submitted 2024-01-06; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Statin eye drop (Experimental): Use of topical atorvastatin eye drop 8 times a day; in addition to eyelid hygiene and artificial tear drops (8 weeks)
  Interventions: Drug: Statin eye drop
- Control (Placebo Comparator): Use of topical eye drops as a placebo same as intervention group but without active ingredient of atorvastatin 8 times a day; in addition to eyelid hygiene and artificial tear drops (8 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Statin eye drop — Use of topical atorvastatin eye 8 times a day; in addition to eyelid hygiene and artificial tear drops (8 weeks)
  Other Names: Tiam Darou
  Arms: Statin eye drop
Drug: Placebo — Use of topical eye drops as a placebo same as intervention group but without active ingredient of atorvastatin 8 times a day; in addition to eyelid hygiene and artificial tear drops (8 weeks)
  Other Names: Tiam Darou
  Arms: Control

SUMMARY:
In the first stage, to evaluate the safety of the topical medication produced by Sina Pharmaceuticals, this medication is experimentally tested on 10 volunteer patients. If no side effects occur, eligible patients are enrolled in the study after examination by a specialist. The second stage is a randomized, double-blind clinical trial, during which selected patients are randomly assigned to the control and intervention groups.

For patients in the intervention group, in addition to standard treatment, including eyelid hygiene and the use of artificial tears, a topical drop of Atorvastatin (50 microM) will be administered, one drop eight times a day in both eyes. In the control group, a placebo will be used in the same manner. The patients will be unaware of their assigned group.

Clinical examinations, including Schirmer's test, tear breakup time, fluorescein staining, and completion of the dry eye syndrome questionnaire and dry eye questionnaire, will be conducted before and after the intervention to assess the level of eye dryness.

ELIGIBILITY:
Inclusion Criteria:

* Age>20 years old
* Dry eye induced by Meibomian gland dysfunction
* Tear break up time less than 10 seconds

Exclusion Criteria:

* Hematologic disorders
* Coagulopathies
* Use of anticoagulant medication
* Use of Peptic ulcer disease
* History of ocular surgeries in the last 3 months
* History of any ocular Malignancies
* History of ocular trauma
* History of statin use

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-01-04 (Estimated); Study Completion 2025-02-04 (Estimated)

PRIMARY OUTCOMES:
Change from tear break up time at week 4 follow up | Baseline and week 4 follow up
  Time taken for the first dry spot to appear on the cornea after a complete blink will be assessed by slit lamp at baseline and week 4 follow up after completion of prescription period (8 week)
Change from tear break up time at week 8 follow up | Baseline and week 8 follow up
  Time taken for the first dry spot to appear on the cornea after a complete blink will be assessed by slit lamp at baseline and week 8 follow up after completion of prescription period (8 week)
Change from tear break up time at week 12 follow up | Baseline and week 12 follow up
  Time taken for the first dry spot to appear on the cornea after a complete blink will be assessed by slit lamp at baseline and week 12 follow up after completion of prescription period (8 week)

SECONDARY OUTCOMES:
Change from Ocular Surface Disease Index at week 4 follow up | Baseline and week 4 follow up
  Ocular Surface Disease Index (OSDI) Questionnaire will be completed by participants at baseline and week 4 follow up after completion of prescription period (8 week)
Change from Ocular Surface Disease Index at week 8 follow up | Baseline and week 8 follow up
  Ocular Surface Disease Index (OSDI) Questionnaire will be completed by participants at baseline and week 8 follow up after completion of prescription period (8 week)
Change from Ocular Surface Disease Index at week 12 follow up | Baseline and week 12 follow up
  Ocular Surface Disease Index (OSDI) Questionnaire will be completed by participants at baseline and week 12 follow up after completion of prescription period (8 week)
Change from dry eye score at week 4 follow up | Baseline and week 4 follow up
  Dry Eye Questionnaire will be completed by participants at baseline and week 4 follow up after completion of prescription period (8 week)
Change from dry eye score at week 8 follow up | Baseline and week 8 follow up
  Dry Eye Questionnaire will be completed by participants at baseline and week 8 follow up after completion of prescription period (8 week)
Change from dry eye score at week 12 follow up | Baseline and week 12 follow up
  Dry Eye Questionnaire will be completed by participants at baseline and week 12 follow up after completion of prescription period (8 week)

CONTACTS AND LOCATIONS:
Overall Officials: Kiana Hassanpour, Principal Investigator — Ophthalmic Research Center
Locations (1):
- Ophthalmic Research Center, Tehran, Iran